

## PARTICIPANT CONSENT FORM

**Study title** - Comparing the effectiveness of computer-aided-design computer-aided-manufacture (CAD/CAM) insoles manufactured from foam-box cast vs direct scan on patient reported outcome measures: A double-blinded, randomised controlled trial.

**Short title** – Comparing clinical outcomes using two insole manufacture techniques.

| Unique | participant number: I | nitials: | Month/Year of Birth: | |
|---|---|---|---|---|
| | | | ir | Participant<br>nitial each point |
| 1. | I confirm that I have read and under (version 2.0) for the above study and understand that my participation is volumithout my medical care or legal rights | d have had the oppor untary and that I am fre | tunity to ask questions. | I |
| 2. | I give permission for the research team to use my medical records for the purpose of this study | | | f |
| 3. | I understand that my medical records may be looked at by authorised individuals from the Sponsor for the study, the UK Regulatory Authority or the Independent Ethics Committee in order to check that the study is being carried out correctly. I give permission, provided that strict confidentiality is maintained, for these bodies to have access to my medical records for the above study and any further research that may be conducted in relation to it. | | | S<br>S<br>S |
| 4. | I understand that even if I withdraw from will be used in the analysis of the reconsent for this. I understand that my | sults of the trial, unle | ss I specifically withdraw | |
| 5. | I consent to the storage including election of this study. I understand that any is strictly confidential and that no personation or other publications. | information that could | l identify me will be kept | t |
| 6. | I agree for my anonymised data to be<br>NHS Greater Glasgow and Clyde and<br>undertaking this research. | | | |
| 7. | I agree to be contacted about future o | pportunities to particip | ate in research | |
| 8. | I agree to take part in the study. | | | |

Short title: Comparing clinical outcomes using two insole manufacture techniques IRAS Project ID: 317502

Version Number: 2.0 08.09.2022

| Name of the participant | Participant's signature and the date the participant signed the consent form |
|---|---|
| Name of the Investigator taking written consent | Investigator's signature and date the Investigator signed the consent form |
| Original to be retained and filed in | the site file. 1 copy to participant, 1 copy to be filed in participant's notes |